CLINICAL TRIAL: NCT05171244
Title: Use of Immersive Virtual Reality to Train the Multisensory Processing Capacities of Children Aged 8 to 16 Years-old With an Autism Spectrum Disorder: Single-center Randomized Pilot Study in Parallel Groups - SEVIRE. (Sensory Virtual Reality)
Acronym: SEVIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DR200078
Record Dates: First submitted 2021-11-18; First posted 2021-12-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Single-center Randomized Pilot Study in Parallel Groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Behavioral: virtual reality training; Behavioral: usual care
- Control group (Sham Comparator)
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: virtual reality training — training of multisensory processing capacities in virtual reality in addition to usual program of interventions in usual care
  Arms: Experimental group
Behavioral: usual care — usual program of interventions in usual care

SUMMARY:
Autism Spectrum Disorder (ASD) is defined as a neurodevelopmental disorder that affects the functioning and development of social communication (DSM5 - 2013). ASD causes particularities in sensory treatments (auditory, visual), qualified as uni-modal. Added to this, there is difficulties to deal with prevailing stimuli of the environment (pluri-modal) ; parents report the discomfort of their child in this situation with "noisy" behavioral manifestations. Therapeutic social skills programs most often address the subject's lack of adjustment to their environment through understanding social rules and codes and cognitive treatment of situations.

Thus, in order to relieve the sensory modulation disorders which can be the cause of social adjustment difficulties, it's propose to exercise the sensory habituation of children with ASD thanks to virtual reality scenarios restored in 3D immersion booth (the CAVE). The child will be exposed to multimodal stimulation during immersion sessions reproducing the conditions of an ecological environment. A therapist will accompany the child in the CAVE throughout the session.

The investigators hypothesize that regular and repeated exposure to a simulated environment in the CAVE can improve multisensory treatment capacities and have a beneficial effect on the autonomy of children and adolescents with ASD in everyday situations.

ELIGIBILITY:
Inclusion Criteria:

* Child / adolescent aged 8 to 16 years, diagnosed with ASD (DSM-5, ADOS, ADI-R criteria).
* Without intellectual delay (QNV> 70, WISC-IV or V, WAIS-III or IV).
* Benefiting from a treatment program at the University Center for Child Psychiatry (CHRU Bretonneau-Tours).
* Schooled in the ordinary school context (primary school, middle school, high school, ULIS).
* Having expressed their agreement to participate in the study.

  * Whose parents or legal representatives have signed written consent.
  * Whose parents or legal representatives are affiliated or beneficiaries of a social security scheme.

Exclusion Criteria:

* Neuromotor disorders.
* Uncorrected visual disorders.
* Hearing impairment.
* Known epilepsy.
* Anxiety syndromes identified.
* Hyper ADD / H type activity.
* Treatment with methylphenidate. - Rare genetic syndrome.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Vineland Adaptive Behavior Scales II (VABS II) score | Baseline, week 15 (after training), 6 months after training
  Behavioral scale VABS II is a test for assessing autonomy of child/adolescent in everyday life. From 0 to 108, higher is the score, more independent the person is in the rated field.

SECONDARY OUTCOMES:
Measures of autistic behaviour by Autism Behavior Rating Scale (ECA2) | Baseline, week 15 (after training), 6 months after training
  ECA2 provides an assessment of the current extent of the child's behavioral characteristics. Scale reportes a score from 0 to 4, 5 levels according to the current importance of these behaviors (0 :absent - 4 :very serious)
Measures of autistic behaviour by Autism Behavior Rating Scale for Parents (ECA2P) | baseline, week 15 (after training), 6 months after training
  ECA2P provides an assessment of the current extent of the child's behavioral characteristics. Scale reportes a score from 0 to 4, 5 levels according to the current importance of these behaviors (0 :absent - 4 :very serious)
Measures of autistic behaviour by Dunn sensory profile | Baseline, week 15 (after training), 6 months after training
  Dunn sensory profile is completed by the parents. From 0 to 110, higher is the score more important is the comportement
Measures of autistic behaviour by Vineland Adaptive Behavior Scales II (VABS II) | Baseline, week 15 (after training), 6 months after training
  VABS-II provides an assessment of problematic behaviour. From 0 to 108, higher is the score, more independent the person is in the rated field.
Cognitive rigidity measure | Baseline, week 15 (after training), 6 months after training
  Neuropsycological tests
Cognitive rigidity measure by rating scale of repeated en restricted behaviours (EC2R) | Baseline, week 15 (after training), 6 months after training
  Evaluation of intensity scores for signs of stereotyped and repetitive activity on the EC2R.Factor sensory-motor stereotypies is evaluated by a score from 0 to 44. Factor reaction to change and modulating insufficiency factor are evaluated by a score from 0 to 28. Factor restricted behaviors is evaluated by a score from 0 to 32. Higher is the score more important is the severity.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Le Centre universitaire de pédopsychiatrie, Tours
  - Pedopsychiatry, University Hospital, Tours, Tours